CLINICAL TRIAL: NCT00005085
Title: A Phase II Study of Rebeccamycin Analogue NSC 655649 in Patients With Metastatic Colorectal Cancer (IMT Codes 23988, 23989, 23993)
Brief Title: Rebeccamycin Analog in Treating Patients With Metastatic or Locally Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067695; AECM-T99-0109; NCI-T99-0109
Record Dates: First submitted 2000-04-06; First posted 2004-03-16 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2002-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — becatecarin

ARMS (1):
- Arm I (Experimental): Patients receive rebeccamycin analogue IV once on day 1. Treatment repeats every 21 days for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.
  Interventions: Drug: becatecarin

INTERVENTIONS:
Drug: becatecarin

SUMMARY:
Phase II trial to study the effectiveness of rebeccamycin analog in treating patients who have metastatic or locally recurrent colorectal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate of patients with metastatic or locally recurrent colorectal cancer treated with rebeccamycin analogue.

II. Determine the toxicity of this regimen in this patient population. III. Determine the effect of this regimen on progression-free and overall survival in these patients.

OUTLINE: This is a multicenter study.

Patients receive rebeccamycin analogue IV once on day 1. Treatment repeats every 21 days for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or locally recurrent adenocarcinoma of the colon or rectum
* No curable stage of disease
* At least 1 unidimensionally measurable lesion
* At 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No tumor lesions in previously irradiated area except clearly measurable lesion documented histologically to be consistent with recurrent tumor in previously irradiated bed within pelvis
* The following are considered nonmeasurable disease:

  * Bone lesions Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Inflammatory breast disease
  * Lymphangitis cutis/pulmonis
  * Abdominal masses not confirmed and followed by imaging techniques
  * Cystic lesions
  * No known brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2 OR Karnofsky 60-100%
* Life expectancy: More than 12 weeks
* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* Eligible for placement of a central venous catheter
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to rebeccamycin analogue
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No concurrent prophylactic growth factors (e.g., epoetin alfa) except for clinically defined indication (e.g., filgrastim (G-CSF) for febrile neutropenia)
* At least 4 weeks since prior chemotherapy (e.g., fluorouracil, oral fluoropyrimidines, irinotecan, or oxaliplatin) (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* No concurrent hormones except for clinically defined indication
* At least 4 weeks since prior radiotherapy (including to bony sites, whole pelvis, lung, liver, or spinal cord/brain) and recovered
* No prior total dose of radiotherapy more than 7,000 cGy
* No prior radiotherapy to 40% or more of total bone marrow
* No prior radiotherapy to only site of measurable disease
* No concurrent radiotherapy
* Recovered from prior therapy 1 prior adjuvant treatment allowed 1 prior treatment for advanced disease allowed
* At least 4 weeks since prior investigational agents
* No other concurrent investigational antineoplastic drugs
* No other concurrent investigational agents
* No concurrent commercial agents for colorectal cancer
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-02; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Atlanta Cancer Care, Atlanta, Georgia
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York